CLINICAL TRIAL: NCT03556540
Title: Influence of Exercise in Patients With Chronic Kidney Disease During Hemodialysis on Cardiac Autonomic Modulation, Function e Quality of Life
Brief Title: Influence of Exercise in Patients With Chronic Kidney Disease During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, DOCTOR, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2.075.500
Record Dates: First submitted 2017-06-29; First posted 2018-06-14 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease; Hemodialysis; Exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Each participant will perform 30 minutes of aerobic on cycle ergometer. The exercise will begin 30 minutes after the start of hemodialysis performed three times a week for three months.
  The sessions will be divided into heating, conditioning and cooling. In the warm-up phase 5 minutes of exercise will be performed between 60-70% of maximal heart rate, with Borg between 1 and 2. In the conditioning phase, 20 minutes of moderate exercise will be performed, with HR between 70-80% And Borg (modified) between 3 and 4. And the quench phase will be 5 min, with FC between 60-70% of the maximum and Borg (modified) between 1 and 2.
  Exercise will be discontinued if the participant has a systolic pressure above 180mmHg, a diastolic pressure above 95mmHg, a 20% change in heart rate, a saturation of less than 88%, physical exhaustion, chest pain, dyspnoea, dizziness and fatigue of the exercised limbs .
Who Masked: Participant, Investigator
Masking Description: Volunteers will not know that there are two groups. Evaluators will not know which groups the volunteers belong to when evaluating the variables.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The volunteers without performing exercise during hemodialysis. Autonomic heart rate modulation, quality of life, physical fitness and safety level of exercise will be evaluated.
  Interventions: Other: physical exercise
- Experimental (Experimental): The volunteers will perform physical exercise during hemodialysis. Autonomic heart rate modulation, quality of life, physical fitness and safety level of exercise will be evaluated.
  Interventions: Other: physical exercise

INTERVENTIONS:
Other: physical exercise — Each participant will perform 30 minutes of aerobic physical activity, using cycle ergometer. The exercise will begin 30 minutes after the start of hemodialysis.

SUMMARY:
Introduction: Chronic Renal Failure affects a large part of the world population, being characterized by irreversible renal tissue damage, resulting in systemic disturbances that negatively affect the patient's life. The most commonly used treatment is hemodialysis, which also has certain deleterious effects, so it is necessary to look for therapies that minimize these complications. Objective: To analyze the influence of physical exercise during hemodialysis on the autonomic heart rate modulation, quality of life and physical functional ability in individuals with Chronic Renal Failure at Hospital das Clínicas Gaspar Vianna. Method: The intervention consists on performing aerobic exercise during hemodialysis. For the evaluation will be applied the KDQOL-SF ™ 1.3 questionnaire, for quality of life; 6-Minute Walk Test for physical functional ability; and cardiofrequencimeter for the autonomic heart rate modulation. Data will be stored in Microsoft Excel® spreadsheets, it will also be used for making graphs and tables. Statistical analysis will be performed in the Bioestat 5.3® program and the choice of tests will depend on the distribution and homogeneity of the data.

DETAILED DESCRIPTION:
This is a randomized, prospective and quantitative clinical trial, whose patients will be selected after analysis of the inclusion and exclusion criteria, which will be performed in the Hemodialysis sector of the State Public Foundation Gaspar Vianna Clinical Hospital.

The target population of this study will consist of individuals with chronic renal failure undergoing hemodialysis. The volunteers of the study will be randomly randomized by a blind researcher who does not know the protocol, groups or volunteers that will be inserted in the study, being allocated in Control Group and Experimental Group.

The sample calculation was performed using the GraphPad StatMate application, version 1.01, with a significance of 5% and a test power of 80%, being used as reference the number of cases found in the literature, being determined that 20 volunteers will be included in the study With chronic kidney disease and who undergo hemodialysis treatment.

In the study, individuals who attend the Monteiro Leite Hemodialysis Center, aged 40 to 70 years, undergoing hemodialysis, only in the FPEHCGV, 3 times a week with a minimum of 6 months of hemodialysis.

Will be excluded from the research, individuals who are hospitalized at the Gaspar Vianna Clinic Hospital or that during the application of the protocol are hospitalized, have osteomioarticular diseases that prevent the proposed exercise, patients who use drugs that influence the heart rhythm , Patients with values of less than 24 points in the evaluation of the mini state of mental assessment, patients with a pacemaker installed, patients who underwent previous cardiac surgery less than six months, patients with a body mass index greater than 30 / kg / m2 .

For the data collection will be used: Polarimeter of the brand POLAR®, model RS800CX (Polar Electro TM, Kempele, Finland); Premium® Aneroid Sphygmomanometer and Premium® Brand Stethoscope, Rappaport Model (Wenzhou Instruments Co; China); Nonin Pulse Oximeter, KDQOL - SF ™ 1.3 Scale and Modified Borg Scale (CR10). Samples will be collected in the control and experimental groups before the start of the protocol, 1 month after protocol initiation, at the end of the protocol and 1 month after the end of the protocol.

For the evaluation of the autonomic modulation of the HR will be used the analysis of the variability of the same, at the moment of the evaluation, after one month of intervention, in the second month and at the end of the collection. The collections will be performed between 8:00 a.m. to 12:00 p.m. and 3:00 p.m. to 7:00 p.m., in order to minimize influences of the circadian cycle on the variability of the HR.

During the evaluation, respiratory rate and blood pressure will be monitored in order to discard their influence on heart rate variability.

At collection, the patients will be positioned first in prone and then supine and finally in standing position. For each analysis, they will be kept in rest for 10 minutes - at each position - allowing the stabilization of vital signs. Next, the HR and the iR-R will be recorded, with a duration of 10 minutes, and the patient will be advised not to perform movements and not to talk during the collection period.

The recording of HRV will be performed by means of a POLAR® brand, RS800CX (Polar Electro ™, Kempele, Finland) cardiofrequency meter, where the HR signal will be captured by a tape with the signal receiver, placed in the thorax of the Patient at the time of the xiphoid process of the sternum.

The transfer of the data recorded by the frequencymeter will be evaluated for the Polar ProTrainer Software (Polar Electro OY, Kempele, Finland) through an infrared signal emitting interface, where it will be stored and subsequently exported in .txt format so that later , Is analyzed in the program Kubios HRV 2.2 (MATLAB, Kuopio, Finland) and saved in the computer with the collection time.

For the analysis, there will be a selection of a five-minute stretch containing the highest signal stability, discarding the initial 30 seconds and the final 30 seconds of collection, provided that it comprises at least 5 minutes or 256 points.

The analysis of the variables in the time domain will be: square root of the square mean of the differences between adjacent normal RR intervals (rMSSD), standard deviation of all normal RR intervals recorded in a time interval (SDNN), and variables in the domain of the Frequency: low frequency spectral component (BF), high frequency spectral component (AF), BF / AF ratio and nonlinear variables: Poincaré plot width (SD1), and Shannon entropy.

It will be evaluated by the 6-Minute Walk Test. It is performed from the placement of 2 cones, one at each end of a 30-meter course. The maximum distance covered by the patient is evaluated in 6 minutes, with walking rhythm respecting its limits, and can not run.

Heart and respiratory rate, blood pressure, shortness of breath, fatigue in the legs from the Borg scale, and blood oxygenation should be checked before and after the test. The following variables were evaluated: heart rate, O2 saturation and Borg scale in the third minute of the test.

For the evaluation of the quality of life, the KDQOL - SF ™ 1.3 Questionnaire will be used, which is an instrument of easy administration and comprehension that has already been validated in Brazil. Its application will take place as follows: the questionnaire will be delivered to the participant and the doubts will be solved, thus enabling the individual to fill out the instrument properly. If the individual is not literate, the evaluators will only assist in reading the questionnaire and answering questions.

The level of safety will be evaluated by constant monitoring of cardiorespiratory variables, such as heart rate, oxygen pulse saturation, respiratory rate and blood pressure, which will be verified and monitored throughout the duration of the technique.

The determination of the protocol was based on a previous study carried out. After randomization of the groups the volunteers of the experimental group will carry out a proposed protocol.

Each participant will perform 30 minutes of aerobic physical activity, using cycle ergometer (Physycal, Londrina, Brazil). The exercise will begin 30 minutes after the start of hemodialysis, and will be performed three times a week for three months.

Before starting the session, a sphygmomanometer, an oximeter and a heart rate monitor will be placed during the procedure. By control, blood pressure, heart rate, peripheral saturation and the Borg Scale will be evaluated every 5 minutes. The heart rate variability will be evaluated every day between the hours of 8:00 a.m. to 12:00 a.m., in rest of 10 minutes in the positions of dorsal decubitus, sedestation and standing.

The sessions will be divided into 3 phases: heating, conditioning and cooling. In the warm-up phase 5 minutes of exercise will be performed between 60-70% of maximal heart rate, with Borg (modified) between 1 and 2. In the conditioning phase, 20 minutes of moderate exercise will be performed, with HR between 70-80% And Borg (modified) between 3 and 4. And the quench phase will be 5 min, with FC between 60-70% of the maximum and Borg (modified) between 1 and 2. The maintenance of the parameters will be regulated by the speed of realization of the exercise.

Exercise will be discontinued if the participant has a systolic pressure above 180mmHg, a diastolic pressure above 95mmHg, a 20% change in heart rate, a saturation of less than 88%, physical exhaustion, chest pain, dyspnoea, dizziness and fatigue of the exercised limbs.

ELIGIBILITY:
Inclusion Criteria:

* Will be included in the research patients with chronic kidney disease, aged 40 to 70 years, undergoing hemodialysis

Exclusion Criteria:

* Will be excluded from the research, individuals who are hospitalized or that during the application of the protocol are hospitalized, have osteomioarticular diseases that prevent the proposed exercise, patients who use drugs that influence the heart rhythm , Patients with values of less than 24 points in the evaluation of the mini state of mental assessment, patients with a pacemaker installed, patients who underwent previous cardiac surgery less than six months, patients with a body mass index greater than 30 / kg / m2 .

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic modulation by heart rate variability | Change from baseline heart rate variability at 3 months
  Cardiac Autonomic modulation was avaliated by Heart rate variability with Polar RS800CX
Quality of life by Kidney Disease and Quality of Life Short Form 1.3 scale | Change from baseline quality of life at 3 months
  Avaliable by Kidney Disease and Quality of Life Short Form 1.3 scale, this scale was divided in 4 domains: Your Health, Kidney Disease, Effects of kidney disease on your daily life and Satisfaction with treatment, each item is put on 0 (worst) to 100 range (better)
Functional capacity by 6-minute walk test | Change from baseline 6-minute walk test at 3 months
  avaliable by 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Rocha, Doctor, Principal Investigator — C
Locations (1):
- Hospital de Clínicas Gaspar Viana, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu YM, Chung YC, Chang JS, Yeh ML. Effects of aerobic exercise during hemodialysis on physical functional performance and depression. Biol Res Nurs. 2015 Mar;17(2):214-21. doi: 10.1177/1099800414539548. Epub 2014 Jul 15. PMID 25027035
- [Result] National Kidney Foundation. KDOQI Clinical Practice Guideline for Hemodialysis Adequacy: 2015 update. Am J Kidney Dis. 2015 Nov;66(5):884-930. doi: 10.1053/j.ajkd.2015.07.015. PMID 26498416
- [Result] Martin-Alemany G, Valdez-Ortiz R, Olvera-Soto G, Gomez-Guerrero I, Aguire-Esquivel G, Cantu-Quintanilla G, Lopez-Alvarenga JC, Miranda-Alatriste P, Espinosa-Cuevas A. The effects of resistance exercise and oral nutritional supplementation during hemodialysis on indicators of nutritional status and quality of life. Nephrol Dial Transplant. 2016 Oct;31(10):1712-20. doi: 10.1093/ndt/gfw297. Epub 2016 Aug 10. PMID 27510532
- [Result] Painter P, Carlson L, Carey S, Paul SM, Myll J. Physical functioning and health-related quality-of-life changes with exercise training in hemodialysis patients. Am J Kidney Dis. 2000 Mar;35(3):482-92. doi: 10.1016/s0272-6386(00)70202-2. PMID 10692275